CLINICAL TRIAL: NCT01332305
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Response Study to Assess the Efficacy, Safety, and Pharmacokinetics of XP13512 (GSK1838262) in Patients With Restless Legs Syndrome
Brief Title: Dose-Response and Pharmacokinetics of Gabapentin Enacarbil (GEn [XP13512 / GSK1838262]) in Restless Legs Syndrome
Acronym: XP081
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: XenoPort, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 111462
Record Dates: First submitted 2011-04-07; First posted 2011-04-11 (Estimated); Results first posted 2011-05-26 (Estimated); Last update posted 2013-07-22 (Estimated); Status verified 2011-05

CONDITIONS: Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome | interventions — 1-(((alpha-isobutanoyloxyethoxy)carbonyl)aminomethyl)-1-cyclohexaneacetic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- GEn (XP13512/GSK1838262) 600 mg (Experimental): GEn (XP13512/GSK1838262) 600 mg
  Interventions: Drug: GEn (XP13512/GSK1838262)
- GEn (XP13512/GSK1838262) 1200 mg (Experimental): GEn (XP13512/GSK1838262) 1200 mg
  Interventions: Drug: GEn (XP13512/GSK1838262)
- GEn (XP13512/GSK1838262) 1800 mg (Experimental): GEn (XP13512/GSK1838262) 1800 mg
  Interventions: Drug: GEn (XP13512/GSK1838262)
- GEn (XP13512/GSK1838262) 2400 mg (Experimental): GEn (XP13512/GSK1838262) 2400 mg
  Interventions: Drug: GEn (XP13512/GSK1838262)
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GEn (XP13512/GSK1838262) — Double-Blind Treatment Phase: 600 mg GEn (XP13512) orally, once daily for 3 days followed by 600 or 1200 mg on days 4-6, followed by 600 or 1200 or 1800 mg on days 7-9, followed by 600 or 1200 or 1800 or 2400 mg on days 10-84. Double-Blind Taper Phase: 600 or 1200 or 1800 mg GEn (XP13512) orally, once daily on days 85-86, followed by 600 mg or 1200 mg on days 87-88, followed by 600 mg on days 89-91
  Other Names: XP13512; GSK1838262
  Arms: GEn (XP13512/GSK1838262) 1200 mg; GEn (XP13512/GSK1838262) 1800 mg; GEn (XP13512/GSK1838262) 2400 mg; GEn (XP13512/GSK1838262) 600 mg
Drug: Placebo — Placebo orally once daily
  Arms: Placebo

SUMMARY:
The objective of the study was to generate the data necessary to determine the gabapentin exposure produced by 4 dose levels of GEn (600 mg, 1200 mg, 1800 mg, and 2400 mg) or placebo, and the corresponding relief of symptoms in subjects with Restless Legs Syndrome (RLS).

DETAILED DESCRIPTION:
This was a multicenter, randomized, double blind, placebo controlled, parallel group study, comparing 4 doses of GEn (XP13512) with placebo given once daily to subjects with RLS. Eligible subjects were randomized in equal numbers into 1 of 5 treatment groups (GEn 600 mg, 1200 mg, 1800 mg, or 2400 mg or placebo) for 12 weeks of treatment. Data from this study will be utilized as part of a larger pharmacokinetic (PK) pharmacodynamic (PD) analysis of data from several studies (XP084/RXP111495) that are part of the GEn RLS clinical development program. Safety and tolerability were also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Men or women at least 18 years of age
* RLS, based on the IRLSSG Diagnostic Criteria
* History of RLS symptoms occurring at least 15 nights in the month prior to Screening or, if on RLS treatment, this frequency of symptoms must have been applicable prior to start of treatment
* Documented RLS symptoms for at least 4 of the 7 consecutive evenings/nights
* Total RLS severity score of 15 or greater on the IRLS Rating Scale
* If taking dopamine agonists, gabapentin, or other treatments for RLS (e.g., opioids, benzodiazepines) medications must have been discontinued at least 2 weeks prior to Screening;
* If taking any prescription medication, therapy must have been stabilized for at least 3 months prior to Screening with no anticipated changes for the duration of the study;
* Body Mass Index (BMI) of 34 or below
* estimated creatinine clearance of at least 60 mL/min

Exclusion Criteria:

* a sleep disorder (e.g., sleep apnea) that may significantly affect the assessment of RLS
* history of RLS symptom augmentation or end of dose rebound with previous dopamine agonist treatment
* neurologic disease or movement disorder (e.g., diabetic neuropathy, Parkinson's disease, multiple sclerosis, dyskinesias, and dystonias);
* other clinically significant or unstable medical condition or conditions which could affect RLS treatment efficacy assessments
* serum ferritin level below 20 ng/mL
* currently suffering from moderate or severe depression using the Diagnostic and Statistical Manual of Mental Disorders and Treatment IV (DSM IV TR)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2007-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Dallas, Texas, United States

REFERENCES:
- [Derived] Ahmed M, Hays R, Steven Poceta J, Jaros MJ, Kim R, Shang G. Effect of Gabapentin Enacarbil on Individual Items of the International Restless Legs Study Group Rating Scale and Post-sleep Questionnaire in Adults with Moderate-to-Severe Primary Restless Legs Syndrome: Pooled Analysis of 3 Randomized Trials. Clin Ther. 2016 Jul;38(7):1726-1737.e1. doi: 10.1016/j.clinthera.2016.05.008. Epub 2016 Jun 7. PMID 27288210
- [Derived] Avidan AY, Lee D, Park M, Jaros MJ, Shang G, Kim R. The Effect of Gabapentin Enacarbil on Quality of Life and Mood Outcomes in a Pooled Population of Adult Patients with Moderate-to-Severe Primary Restless Legs Syndrome. CNS Drugs. 2016 Apr;30(4):305-16. doi: 10.1007/s40263-016-0329-4. PMID 27067343
- [Derived] Ondo WG, Hermanowicz N, Borreguero DG, Jaros MJ, Kim R, Shang G. Effect of prior exposure to dopamine agonists on treatment with gabapentin enacarbil in adults with moderate-to-severe primary restless legs syndrome: pooled analyses from 3 randomized trials. J Clin Mov Disord. 2015 Mar 30;2:9. doi: 10.1186/s40734-015-0018-3. eCollection 2015. PMID 26788345
- [Derived] Lal R, Ellenbogen A, Chen D, Zomorodi K, Atluri H, Luo W, Tovera J, Hurt J, Bonzo D, Lassauzet ML, Vu A, Cundy KC. A randomized, double-blind, placebo-controlled, dose-response study to assess the pharmacokinetics, efficacy, and safety of gabapentin enacarbil in subjects with restless legs syndrome. Clin Neuropharmacol. 2012 Jul-Aug;35(4):165-73. doi: 10.1097/WNF.0b013e318259eac8. PMID 22664749

RESULTS

PARTICIPANT FLOW:
Groups:
- GEn Placebo: Oral placebo tablet taken once daily. Days 1 to 3: one placebo tablet. Days 4 to 6: two placebo tablets. Days 7 to 9: three placebo tablets. Days 10 to 84: four placebo tablets. On Day 85, participants entered a 7-day Taper Period. Days 85 to 86: three placebo tablets. Days 87 to 88: two placebo tablets. Days 89 to 91: one placebo tablet.
- GEn 600 mg: Gabapentin enacarbil (GEn) (XP13512/GSK1838262) 600 milligrams (mg) taken orally once a day for 12 weeks. Days 1 to 3: one extended release (ER) tablet (600 mg GEn). Days 4 to 6: one ER tablet (600 mg GEn) and one placebo tablet. Days 8 to 10: one ER tablet (600 mg GEn) and two placebo tablets. Days 10 to 84: one ER tablet (600 mg GEn) and three placebo tablets. On Day 85, participants entered a 7-day Taper Period. Days 85 to 86: three placebo tablets. Days 87 to 88: two placebo tablets. Days 89 to 91: one placebo tablet.
- GEn 1200 mg: Oral GEn 1200 mg taken once daily. Days 1 to 3: one ER tablet (600 mg GEn). Days 4 to 6: two ER tablets (1200 mg GEn). Days 8 to 10: two ER tablets (1200 mg GEn) and one placebo tablet. Days 10 to 84: two ER tablets (1200 mg GEn) and two placebo tablets. On Day 85, participants entered a 7-day Taper Period. Days 85 to 86: one ER tablet (600 mg GEn) and two placebo tablets. Days 87 to 88: two placebo tablets. Days 89 to 91: one placebo tablet.
- GEn 1800 mg: Oral GEn 1800 mg taken once daily. Days 1 to 3: one ER tablet (600 mg GEn). Days 4 to 6: two ER tablets (1200 mg GEn). Days 8 to 10: three ER tablets (1800 mg GEn). Days 10 to 84: three ER tablets (1800 mg GEn) and one placebo tablet. On Day 85, participants entered a 7-day Taper Period. Days 85 to 86: two ER tablets (1200 mg GEn) and one placebo tablet. Days 87 to 88: one ER tablet (600 mg) and one placebo tablet. Days 89 to 91: one placebo tablet.
- GEn 2400 mg: Oral GEn 1200 mg taken once daily. Days 1 to 3: one ER tablet (600 mg GEn). Days 4 to 6: two ER tablets (1200 mg GEn). Days 8 to 10: three ER tablets (1800 mg GEn). Days 10 to 84: four ER tablets (2400 mg GEn). On Day 85, participants entered a 7-day Taper Period. Days 85 to 86: three ER tablets (1800 mg GEn). Days 87 to 88: two ER tablets (1200 mg). Days 89 to 91: one ER (600 mg) tablet.
Period: Overall Study
Arm/Group | GEn Placebo | GEn 600 mg | GEn 1200 mg | GEn 1800 mg | GEn 2400 mg
Started | 41 | 48 | 45 | 38 | 45
Completed | 31 | 34 | 31 | 30 | 33
Not Completed | 10 | 14 | 14 | 8 | 12
Not completed — Adverse Event | 1 | 4 | 6 | 3 | 5
Not completed — Withdrawal by Subject | 6 | 5 | 4 | 1 | 0
Not completed — Lost to Follow-up | 0 | 2 | 3 | 2 | 3
Not completed — Protocol Violation | 1 | 2 | 1 | 0 | 3
Not completed — Withdrawal by Sponsor | 1 | 0 | 0 | 1 | 1
Not completed — Treatment Failure | 1 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GEn Placebo | GEn 600 mg | GEn 1200 mg | GEn 1800 mg | GEn 2400 mg | Total
Number analyzed (Participants) | 41 | 48 | 45 | 38 | 45 | 217
Age Continuous [Mean (Standard Deviation); unit: Years] | 47.1 (11.16) | 47.3 (12.78) | 49.8 (11.51) | 50.2 (13.79) | 45.9 (13.93) | 48.0 (12.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 31 | 23 | 27 | 29 | 139
  Male | 12 | 17 | 22 | 11 | 16 | 78
Race/Ethnicity, Customized [Number; unit: participants] — There was one participant in the GEn 2400 mg arm who was categorized in more than one race.
  participants
    White or Caucasian | 39 | 48 | 44 | 35 | 42 | 208
    Black or African American | 1 | 0 | 1 | 2 | 2 | 6
    American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1 | 2
    Asian | 0 | 0 | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Mean Css, Max and Css, Min
Description: Css, max is defined as the maximum or "peak" concentration of a drug observed after multiple administration, at steady state. Css, max is one of the parameters of particular use in estimating the bioavailability of drugs, by measuring the total amount of drug absorbed. Css, min is defined as the minimum concentration of a drug observed after its administration, in steady state. ng, nanograms; PK, pharmacokinetic; W, week; BLQ, below limit of quantitation.
Time Frame: Weeks 4 and 12
Population: Safety Population: all participants (par.) who were randomized and received at least one (or any portion of a) dose of study drug. Population was analyzed as randomized. Placebo par. had no exposure to GEn and were not included in the PK assessments. Of par. who completed the study, some were not included at W12 (sample not taken or BLQ).
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/ml)
Arm/Group | GEn Placebo | GEn 600 mg | GEn 1200 mg | GEn 1800 mg | GEn 2400 mg
Number analyzed (Participants) | 0 | 39 | 33 | 33 | 36
nanograms per milliliter (ng/ml)
  Css, max; Week 4, n=0, 39, 33, 33, 36 |  | 3.86 (1.25) | 7.14 (2.62) | 11.4 (3.54) | 14.0 (4.23)
  Css, max; Week 12, n=0, 32, 30, 30, 31 |  | 4.14 (1.19) | 7.15 (2.76) | 12.0 (3.83) | 13.3 (3.83)
  Css, min; Week 4, n=0, 39, 33, 33, 36 |  | 0.690 (0.359) | 1.37 (0.894) | 1.63 (0.967) | 2.34 (1.78)
  Css, min; Week 12, n=0, 32, 30, 30, 31 |  | 0.600 (0.332) | 1.32 (1.15) | 1.60 (0.994) | 2.41 (1.29)

2. Primary Outcome: Mean Tmax and T1/2
Description: Tmax is defined as the time to the maximum or "peak" concentration of a drug observed after multiple administration. T1/2 is defined as the time to when half of the total amount of a particular substance is eliminated from the body.
Time Frame: Weeks 4 and 12
Population: Safety Population. Placebo participants (par.) were not included in the PK assessments, as they had no exposure to GEn. At W4, there were two par. excluded from the T1/2, as a result of no sample taken or a PK profile not possible. Of par. who completed the study, some were not included at W12 (sample not taken or below limit of quantitation).
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | GEn Placebo | GEn 600 mg | GEn 1200 mg | GEn 1800 mg | GEn 2400 mg
Number analyzed (Participants) | 0 | 39 | 33 | 33 | 36
hours
  Tmax; Week 4, n=0, 39, 33, 33, 36 |  | 8.76 (3.81) | 8.57 (3.16) | 7.61 (2.67) | 8.01 (3.62)
  Tmax; Week 12, n=0, 32, 30, 30, 31 |  | 6.96 (3.76) | 8.72 (3.68) | 8.00 (2.58) | 8.13 (3.20)
  T1/2; Week 4, n=0, 38, 33, 33, 35 |  | 5.82 (1.46) | 6.67 (1.94) | 5.82 (1.56) | 6.05 (1.11)
  T1/2, Week 12, n=0, 32, 30, 30, 30 |  | 6.27 (1.77) | 6.63 (2.23) | 5.89 (1.36) | 6.09 (1.28)

3. Primary Outcome: Mean AUCss
Description: The area under the plot of plasma concentration of drug against time after drug administration is defined as the area under the curve (AUC). The AUCss is the area under the curve during the steady-state period. The AUCss is of particular use in estimating the bioavailability of drugs, by measuring the extent of absorption. AUCss used concentration data from 0 to 24 hours at steady-state for Weeks 4 and 12.
Time Frame: Weeks 4 and 12
Population: Safety Population. Placebo participants were not included in the PK assessments, as they had no exposure to GEn. Of participants who completed the study, some were not included at Week 12 (sample not taken or below limit of quantitation).
Measure: Mean (Standard Deviation); unit: ng*hour/ml
Arm/Group | GEn Placebo | GEn 600 mg | GEn 1200 mg | GEn 1800 mg | GEn 2400 mg
Number analyzed (Participants) | 0 | 38 | 33 | 33 | 35
ng*hour/ml
  Week 4, n=0, 38, 33, 33, 35 |  | 49.3 (14.8) | 96.1 (30.4) | 141 (41.0) | 176 (53.8)
  Week 12, n=0, 32, 30, 30, 30 |  | 51.4 (16.5) | 95.7 (38.5) | 146 (41.4) | 173 (54.4)

ADVERSE EVENTS:
Time Frame: Treatment-Emergent Adverse Events (TEAEs) were collected from the first dose of randomized study medication through end of taper phase (up to Week 13). Any Serious Adverse Event (SAE) reported up to 30 days after last dose was also reported.
Description: At the end of the follow-up period (30 days after the last day of taper [Day 119]), the study coordinator called participants (+/- 3 day window) who did not enroll in the open-label extension protocol to determine if any SAEs occurred, and the resolution date for any AEs that were ongoing at the end of the study.
Arm/Group | GEn Placebo | GEn 600 mg | GEn 1200 mg | GEn 1800 mg | GEn 2400 mg
Serious Adverse Events (participants affected / at risk) | 1/41 | 0/48 | 1/45 | 0/38 | 1/45
Other Adverse Events (participants affected / at risk) | 21/41 | 24/48 | 33/45 | 25/38 | 42/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GEn Placebo (N=41) | GEn 600 mg (N=48) | GEn 1200 mg (N=45) | GEn 1800 mg (N=38) | GEn 2400 mg (N=45)
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GEn Placebo (N=41) | GEn 600 mg (N=48) | GEn 1200 mg (N=45) | GEn 1800 mg (N=38) | GEn 2400 mg (N=45)
Somnolence (Nervous system disorders) | 2 | 7 | 11 | 10 | 23
Dizziness (Nervous system disorders) | 1 | 10 | 10 | 10 | 18
Headache (Nervous system disorders) | 7 | 2 | 9 | 4 | 6
Nausea (Gastrointestinal disorders) | 5 | 3 | 4 | 3 | 3
Fatigue (General disorders) | 4 | 2 | 4 | 1 | 2
Diarrhea (Gastrointestinal disorders) | 4 | 1 | 3 | 2 | 2
Nasopharyngitis (Infections and infestations) | 3 | 1 | 3 | 3 | 2
Irritability (General disorders) | 2 | 2 | 3 | 2 | 2
Insomnia (Psychiatric disorders) | 1 | 5 | 1 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 2 | 2 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 4 | 2 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 1 | 3 | 0 | 3
Feeling drunk (General disorders) | 0 | 0 | 0 | 3 | 4
Peripheral edema (General disorders) | 1 | 0 | 2 | 1 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2 | 2 | 0
Sedation (Nervous system disorders) | 1 | 0 | 0 | 3 | 3
Constipation (Gastrointestinal disorders) | 0 | 1 | 3 | 2 | 0
Feeling abnormal (General disorders) | 0 | 0 | 2 | 3 | 1
Vision blurred (Eye disorders) | 0 | 0 | 2 | 0 | 4
Disorientation (Psychiatric disorders) | 1 | 0 | 1 | 2 | 1
Non-cardiac chest pain (General disorders) | 1 | 1 | 0 | 0 | 3
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 2 | 1
Depression (Psychiatric disorders) | 0 | 0 | 3 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 3 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 2 | 2
Disturbance in attention (Nervous system disorders) | 0 | 1 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.